CLINICAL TRIAL: NCT02969317
Title: An Open-label Trial to Assess Pharmacokinetics and Safety of Tiotropium + Olodaterol Fixed-dose Combination (5 µg/ 5 µg) Delivered by the RESPIMAT Inhaler After Single and Multiple Dose Treatment in Chinese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Bioavailability of Tiotropium + Olodaterol Fixed-dose Combination (5 μg/ 5 μg) in Chinese COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1237.30
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tiotropium + olodaterol fixed-dose combination (Experimental): Fixed dose combination
  Interventions: Drug: Tiotropium; Drug: Olodaterol

INTERVENTIONS:
Drug: Tiotropium — Fixed dose combination
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO
Drug: Olodaterol — Fixed dose combination
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics of tiotropium + olodaterol fixed-dose combination (FDC) (5 μg/ 5 μg) delivered by the RESPIMAT inhaler after single dose and at steady state in Chinese patients with COPD.

The secondary objective is to assess the safety of tiotropium + olodaterol FDC (5 μg/ 5 μg) delivered by the RESPIMAT inhaler after 3 weeks once daily treatment in Chinese patients with COPD.

ELIGIBILITY:
Inclusion criteria:

* All patients must sign an informed consent consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines and local legislations prior to any study-related procedures, which includes medication washout and restrictions.
* All patients must have a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) and must meet the following spirometric criteria:

Patients must have relatively stable airway obstruction with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) >=30% of predicted normal and <80% of predicted normal (ECSC,; and a postbronchodilator FEV1/ Forced Vital Capacity (FVC)<70% at Visit 1

* Male or female patients, 40 years of age or older.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years.

Patients who have never smoked cigarettes must be excluded.

* Patients must be able to

  * perform technically acceptable pulmonary function tests,
  * maintain medication worksheet records during the study period,
  * perform all other assessments as required in the protocol.
* Patients must be able to inhale medication in a competent manner from the RESPIMAT inhaler and from a metered dose inhaler (MDI).
* Male or female patients. Women of childbearing potential* must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

  * Women of childbearing potential are defined as:

Any female who has experienced menarche and does not meet the criteria for "women not of childbearing potential" as described below.

Women not of childbearing potential are defined as:

Women who are postmenopausal (12 months with no menses without an alternative medical cause) or who are permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion criteria:

* Patients with a significant disease other than Chronic Obstructive Pulmonary Disease (COPD); a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study.
* Patients with a, in the opinion of the investigator, clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an Serum Glutamic Oxaloacetic Transaminase (SGOT) >x 2 Upper Limit of Normal (ULN), Serum Glutamic Pyruvic Transaminase(SGPT) >x 2 ULN, bilirubin >x 2 ULN or creatinine >x 2 ULN will be excluded regardless of clinical condition (a repeat laboratory evaluation will not be conducted in these patients).
* Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma. If a patient has a total blood eosinophil count ≥600/mm3, source documentation is required to verify that the increased eosinophil count is related to a non-asthmatic condition.

Patients with any of the following conditions:

* A diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists).
* A diagnosis of paroxysmal tachycardia (>100 beats per minute) (due to the known class side effect profile of ß2-agonists)
* A history of myocardial infarction within 1 year of screening visit (Visit 1).
* Unstable or life-threatening cardiac arrhythmia.
* Hospitalization for heart failure within the past year.
* Known active tuberculosis.
* A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed).
* A history of life-threatening pulmonary obstruction.
* A history of cystic fibrosis.
* Clinically evident bronchiectasis.
* A history of significant alcohol or drug abuse.
* Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1).
* Patients being treated with oral or patch β-adrenergics.
* Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
* Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
* Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program.
* Patients who have taken an investigational drug within one month or six half lives or within the wash out period (whichever is greater) prior to screening visit (Visit 1).
* Patients with known hypersensitivity to β-adrenergics and/or anticholinergic drugs, benzalkonium chloride (BAC), disodium edentate (EDTA) or any other component of the RESPIMAT inhalation solution.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Women of childbearing potential not using two highly effective methods of birth control*.

Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.

* as per ICH M3: a highly effective method of birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.

* Patients who have previously been allocated in this study or are currently participating in another study.
* Patients who are unable to comply with pulmonary medication restrictions prior to allocation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- West China Hospital, Chengdu, China

REFERENCES:
- [Derived] Wang Z, Tadayasu Y, Hu N, Shu S, Hu C, Luo Z. Pharmacokinetics and safety of tiotropium+olodaterol 5 mug/5 mug fixed-dose combination in Chinese patients with COPD. Pulm Pharmacol Ther. 2020 Aug;63:101944. doi: 10.1016/j.pupt.2020.101944. Epub 2020 Sep 9. PMID 32916296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 patients were entered to receive treatment with tiotropium+olodaterol fixed-dose combination (FDC) 5 microgram / 5 microgram (5 μg / 5 μg). All of the 12 entered patients were treated with trial medication.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Tiotropium+Olodaterol 5 Microgram/5 Microgram: Patients were administered with 2 oral inhalations once daily (AM dosing) via RESPIMAT® inhaler of 2.5 μg per actuation of Tiotropium solution and 2.5 μg per actuation of Olodaterol solution
Period: Overall Study
Arm/Group | Tiotropium+Olodaterol 5 Microgram/5 Microgram
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This set included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Tiotropium+Olodaterol 5 Microgram/5 Microgram
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data were not collected from any participant
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve of Olodaterol in Plasma Over the Time Interval From 0 to 6 Hours After Drug Administration (AUC0-6)
Description: The descriptive statistics of AUC0-6 could not be evaluated. Since the plasma concentrations of olodaterol and tiotropium was only quantifiable in less than two-thirds of the patients after 4 hours and 1 hour, respectively, and the descriptive statistics is calculated in case that 2/3 patients of total could be evaluated as defined in Clinical trial Protocol (CTP).
Time Frame: 0:05 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00 (hours:minutes) after drug administration
Population: Pharmacokinetic analysis set (PKS): This set included all patients in the treated set with at least one evaluable PK parameter in the treatment period without important protocol violations related to PK
Groups:
- Tiotropium+Olodaterol FDC 5 mg/5 mg: Patients were administered with 2 oral inhalations once daily (AM dosing) via RESPIMAT® inhaler of 2.5 μg per actuation of Olodaterol solution
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 0

2. Primary Outcome: Time From Dosing to the Maximum Concentration of Olodaterol in Plasma (Tmax)
Description: Tmax, time from dosing to the maximum concentration of olodaterol in plasma after single inhaled administration of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
  detailed sampling time points: 0:05 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00, 143:45, 144:20, 311:45, 312:20, 407:45, 408:20, 431:45, 432:20, 455:45, 456:20(hours:minutes) after drug administration.
Time Frame: Day 1, 7, 14, 18, 19 and 20
Population: PKS (evaluable cases)
Measure: Median (Full Range); unit: Hour [h]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Hour [h] | 0.167 [0.117 to 3.00]

3. Primary Outcome: Maximum Measured Concentration of Olodaterol in Plasma (Cmax)
Description: Cmax, maximum measured concentration of olodaterol in plasma after single inhaled administration of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
  detailed sampling time points: 0:05 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00, 143:45, 144:20, 311:45, 312:20, 407:45, 408:20, 431:45, 432:20, 455:45, 456:20(hours:minutes) after drug administration.
Time Frame: Day 1, 7, 14, 18, 19 and 20
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per millilitre [pg/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Picograms per millilitre [pg/mL] | 1.26 (104)

4. Primary Outcome: Maximum Measured Concentration of Olodaterol in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss, maximum measured concentration of olodaterol in plasma at steady state of olodaterol after multiple dosing at Visit 4 (day 21) of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: Day 21: 0:15 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00, 12:00, 24:00 (hours:minutes) after drug administration
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per millilitre [pg/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Picograms per millilitre [pg/mL] | 2.00 (98.4)

5. Primary Outcome: Pre-dose Concentration of Olodaterol in Plasma at Steady State (Cpre,ss)
Description: Cpre,ss, pre-dose concentration of olodaterol in plasma at steady state after multiple dosing at Day 21 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per millilitre [pg/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 9
Picograms per millilitre [pg/mL] | 0.788 (70.7)

6. Primary Outcome: Area Under the Concentration Time Curve of Olodaterol in Plasma Over the Time Interval From 0 to 6 Hours at Steady State (AUC0-6,ss)
Description: AUC0-6,ss, area under the concentration time curve of olodaterol in plasma over the time interval from 0 to 6 hours at steady state after multiple dosing at Day 21 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: Day 21: 0:15 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00 (hours:minutes) after drug administration
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms*hour per millilitre [pg*h/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Picograms*hour per millilitre [pg*h/mL] | 7.54 (79.7)

7. Primary Outcome: Area Under the Concentration-time Curve of Olodaterol in Plasma at Steady State Over a Uniform Dosing Interval τ at Steady State (AUCτ,ss)
Description: AUCτ,ss, area under the concentration-time curve of olodaterol in plasma at steady state over a uniform dosing interval τ at steady state after multiple dosing at Day 21 is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms*hour per millilitre [pg*h/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 10
Picograms*hour per millilitre [pg*h/mL] | 25.5 (64.7)

8. Primary Outcome: Time From Dosing to the Maximum Concentration of Olodaterol in Plasma at Steady State (Tmax,ss)
Description: Tmax,ss,time from dosing to the maximum concentration of olodaterol in plasma at steady state after multiple dosing at Day 21 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Median (Full Range); unit: Hour [h]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Hour [h] | 2.00 [0.117 to 12.0]

9. Primary Outcome: Accumulation Ratios in Plasma of Olodaterol (RA,Cmax =Cmax,ss/Cmax)
Description: Accumulation ratios in plasma of olodaterol (RA,Cmax =Cmax,ss/Cmax) after multiple dosing at Day 21 is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: Day 1 and Day 21
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Ratio | 1.58 (97.4)

10. Primary Outcome: Accumulation Ratios in Plasma of Olodaterol (RA,AUC =AUC0-6,ss/AUC0-6)
Description: Regarding AUC0-6 and RA,AUC0-6, the descriptive statistics of AUC0-6 could not be evaluated. Since the plasma concentrations of olodaterol and tiotropium was only quantifiable in less than two-thirds of the patients after 4 hours and 1 hour, respectively, and the descriptive statistics is calculated in case that 2/3 patients of total could be evaluated as defined in Clinical trial Protocol (CTP). And RA,AUC0-6 is the ratio of AUC0-6,ss to AUC0-6. So, the descriptive RA,AUC0-6 was not calculated either.
Time Frame: Day 1 and Day 21
Population: PKS (evaluable cases)
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 0

11. Primary Outcome: Area Under the Concentration Time Curve of Tiotropium in Plasma Over the Time Interval From 0 to 6 Hours After Drug Administration (AUC0-6)
Description: as for outcome 1
Time Frame: Day 1
Population: PKS (evaluable cases)
Groups:
- Tiotropium+Olodaterol FDC 5 mg/5 mg: Patients were administered with 2 oral inhalations once daily (AM dosing) via RESPIMAT® inhaler of 2.5 μg per actuation of Tiotropium solution
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 0

12. Primary Outcome: Time From Dosing to the Maximum Concentration of Tiotropium in Plasma (Tmax)
Description: Tmax, time from dosing to the maximum concentration of Tiotropium in plasma after single inhaled administration of tiotropium+olodaterol FDC 5 mg/5 mgis presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
  Detailed sampling time points:0:05 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00, 143:45, 144:20, 311:45, 312:20, 407:45, 408:20, 431:45, 432:20, 455:45, 456:20 (hours:minutes) after drug administration
Time Frame: Day 1, 7, 14, 18, 19, 20
Population: PKS (evaluable cases)
Measure: Median (Full Range); unit: Hour [h]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 11
Hour [h] | 0.167 [0.0330 to 2.00]

13. Primary Outcome: Maximum Measured Concentration of Tiotropium in Plasma (Cmax)
Description: Cmax, maximum measured concentration of Tiotropium in plasma after single inhaled administration of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
  Detailed sampling time points:0:05 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00, 143:45, 144:20, 311:45, 312:20, 407:45, 408:20, 431:45, 432:20, 455:45, 456:20 (hours:minutes) after drug administration
Time Frame: Day 1, 7, 14, 18, 19, 20
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per millilitre [pg/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 11
Picograms per millilitre [pg/mL] | 6.12 (83.5)

14. Primary Outcome: Maximum Measured Concentration of Tiotropium in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss, maximum measured concentration of olodaterol in plasma at steady state of Tiotropium after multiple dosing at Visit 4 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per millilitre [pg/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Picograms per millilitre [pg/mL] | 7.65 (112)

15. Primary Outcome: Pre-dose Concentration of Tiotropium in Plasma at Steady State (Cpre,ss)
Description: Cpre,ss, pre-dose concentration of Tiotropium in plasma at steady state after multiple dosing at Visit 4 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per millilitre [pg/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 8
Picograms per millilitre [pg/mL] | 1.90 (30.6)

16. Primary Outcome: Area Under the Concentration Time Curve of Tiotropium in Plasma Over the Time Interval From 0 to 6 Hours at Steady State (AUC0-6,ss)
Description: AUC0-6,ss, area under the concentration time curve of Tiotropium in plasma over the time interval from 0 to 6 hours at steady state after multiple dosing at Visit 4 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: Day 21:0:15 (hours:minutes) before drug administration and 0:02, 0:05, 0:07, 0:10, 0:20, 0:30, 0:40, 1:00, 2:00, 3:00, 4:00, 6:00 (hours:minutes) after drug administration
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms*hour per millilitre [pg*h/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 11
Picograms*hour per millilitre [pg*h/mL] | 22.0 (75.2)

17. Primary Outcome: Area Under the Concentration-time Curve of Tiotropium in Plasma at Steady State Over a Uniform Dosing Interval τ at Steady State (AUCτ,ss)
Description: AUCτ,ss, area under the concentration-time curve of Tiotropium in plasma at steady state over a uniform dosing interval τ at steady state after multiple dosing at Visit 4 is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms*hour per millilitre [pg*h/mL]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 11
Picograms*hour per millilitre [pg*h/mL] | 54.8 (71.8)

18. Primary Outcome: Time From Dosing to the Maximum Concentration of Tiotropium in Plasma at Steady State (Tmax,ss)
Description: Tmax,ss,time from dosing to the maximum concentration of Tiotropium in plasma at steady state after multiple dosing at Visit 4 of tiotropium+olodaterol FDC 5 mg/5 mg is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: as for outcome 4
Population: PKS (evaluable cases)
Measure: Median (Full Range); unit: Hour [h]
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 12
Hour [h] | 0.0830 [0.0330 to 2.0]

19. Primary Outcome: Accumulation Ratios in Plasma of Tiotropium (RA,Cmax =Cmax,ss/Cmax)
Description: Accumulation ratios in plasma of Tiotropium (RA,Cmax =Cmax,ss/Cmax) after multiple dosing at Visit 4 is presented as unadjusted geometric mean (gMean) and geometric coefficient of variation (gCV) (%).
Time Frame: Day 1, 7, 14, 18, 19, 20 and 21
Population: PKS (evaluable cases)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 11
ratio | 1.29 (127)

20. Primary Outcome: Accumulation Ratios in Plasma of Tiotropium (RA,AUC =AUC0-6,ss/AUC0-6)
Description: Regarding AUC0-6 and RA,AUC0-6, the descriptive statistics of AUC0-6 could not be evaluated. Since the plasma concentrations of olodaterol and tiotropium was only quantifiable in less than two-thirds of the patients after 4 hours and 1 hour, respectively, and the descriptive statistics is calculated in case that 2/3 patients of total could be evaluated as defined in CTP. And RA,AUC0-6 is the ratio of AUC0-6,ss to AUC0-6. So, the descriptive RA,AUC0-6 was not calculated either.
Time Frame: Day 1 and Day 21
Population: PKS (evaluable cases)
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first drug administration through the residual effect period (REP) [[REP, defined as 21 days after last trial medication application], until individual patient's end of trial); up to 6 weeks.
Description: All treated subjects (that is, all subjects who received at least 1 dose of trial drug), were included in the safety analysis.
Arm/Group | Tiotropium+Olodaterol FDC 5 mg/5 mg
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium+Olodaterol FDC 5 mg/5 mg (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02969317/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02969317/SAP_001.pdf